CLINICAL TRIAL: NCT05214482
Title: A Phase Ib/II Study of AK112（PD-1 / VEGF Bispecific Antibody） in Combination With AK117（Anti-CD47 Antibody）With or Without Chemotherapy in Advanced Malignant Tumors
Brief Title: A Study of AK112 in Advanced Malignant Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK117-202
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ib (Experimental): Subjects receive AK112 plus AK117 until progression
  Interventions: Drug: AK112; Drug: AK117
- Phase II (Experimental): AK112 + chemotherapy± AK117 until progression; AK117 + chemotherapy;
  Interventions: Drug: AK112; Drug: AK117; Drug: Chemotherapy

INTERVENTIONS:
Drug: AK112 — IV infusion,Specified dose on specified days
Drug: AK117 — IV infusion,Specified dose on specified days
Drug: Chemotherapy — IV infusion,Specified dose on specified days
  Arms: Phase II

SUMMARY:
Phase Ib/II open label, multicenter study to evaluate the efficacy and safety of AK112 (anti-PD-1 and VEGF bispecific antibody) combined with AK117（Anti-CD47 Antibody）with or without chemotherapy in advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Phase Ib:Histologically or cytologically confirmed advanced solid tumor.
5. Phase II:

   cohort 1 : Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic gastric or GEJ adenocarcinoma.

   cohort 2 : Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic Biliary Tract Cancers, including intrahepatic cholangiocarcinoma, extrahepatic bile duct cancer, gallbladder cancer.

   cohort 3 : Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic pancreatic ductal adenocarcinoma.

   cohort 4 : Has a histologically or cytologically confirmed stage IIIB/IIIC (American Joint Committee on Cancer [AJCC] 8th edition) NSCLC that is unresectable and not fit for radical concurrent chemoradiotherapy, or metastatic / recurrent non-squamous NSCLC;Have previously received EGFR-TKI treatment and have progressed on or following.
6. Have at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator.
7. Has adequate organ function.

Exclusion Criteria:

1. Undergone major surgery within 30 days prior to the first dose of study treatment.
2. Active central nervous system (CNS) metastases.
3. History of active autoimmune disease that has required systemic treatment in the past 2 years (i.e.,corticosteroids or immunosuppressive drugs).
4. Active Hepatitis B or Hepatitis C.
5. Received previous immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy and other treatments targeting the mechanism of tumor immunity.
6. History of severe bleeding tendency or coagulation disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 2 years
  Characterization of incidence, severity and abnormal clinically significant laboratory findings of AEs
Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China